CLINICAL TRIAL: NCT02048254
Title: A Randomized Control Trial (RCT) of Using Iodine-125 Brachytherapy Versus Intensity-modulated Radiation Therapy (IMRT) to Treat Inoperable Salivary Gland Cancer
Brief Title: Study of I-125 Brachytherapy Versus Intensity-modulated Radiation Therapy to Treat Inoperable Salivary Gland Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jianguo Zhang, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUCRP201308
Record Dates: First submitted 2014-01-23; First posted 2014-01-29 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Salivary Gland Cancer
Keywords: inoperable salivary gland cancer; brachytherapy; intensity-modulated radiation therapy
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Brachytherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- brachytherapy (Experimental): Iodine-125 radioactive seeds permanent interstitial implantation brachytherapy
  Interventions: Radiation: brachytherapy
- IMRT (Active Comparator): IMRT (intensity-modulated radiation therapy), 6 Millivolt (MV)-x fractionated irradiation, 1 time/day, 5 times a week, till the end. Add up to 33 times.
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: brachytherapy
  Arms: brachytherapy
Radiation: IMRT
  Other Names: intensity-modulated radiation therapy
  Arms: IMRT

SUMMARY:
* To compare the efficacy of Iodine-125 radioactive seeds implantation versus IMRT to treat inoperable salivary gland carcinoma.
* To compare the safety of Iodine-125 radioactive seeds implantation versus IMRT to treat inoperable salivary gland carcinoma.

DETAILED DESCRIPTION:
The target population are those patients with inoperable salivary gland derived primary or recurrent cancer, including local advanced primary salivary gland cancer which could not be resected completely; recurrent salivary gland cancer which could not be resected completely; T3/T4 tumor which could not tolerate surgery due to severe combined disease. The subjects would be divided into Iodine-125 radioactive seeds permanent interstitial implantation brachytherapy and intensity-modulated radiation therapy randomly. During the follow-up period, the efficacy and the safety index would be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients are diagnosed histologically as primary or recurrent salivary gland cancers that may occur in either major salivary glands or minor salivary glands.
* The inoperable circumstance include: Primary or recurrent salivary gland cancers that could not be resected completely or could not get negative incision.
* T3/T4 tumor patients with severe medical comorbidities could not accept the high risk of perioperative complications.
* At least one measurable tumor or focus (according to RESIST 1.1 Standard).
* Karnofsky score> 60.
* Survival time predicted ≥ 3months;
* HGB≥9 g/dL, WBC≥3.0×10^9/L, NEUT≥1.5×10^9/L, platelet count (PLT)≥ 100×10^9/L; TBIL≤1.5 upper limit of normal, Alanine aminotransferase (ALT)/AST≤3 upper limit of normal; Cera≤1.5 upper limit of normal.
* Male or female with fertility in the experiment are willing to take contraceptive measures.

Exclusion Criteria:

* Radioactive therapy history of head and neck.
* Suffering from other malignant tumor in recent five years, except skin basal cell carcinoma or carcinoma in situs of cervix.
* Chemotherapy history.
* Receiving other effective therapy.
* Distant metastases.
* Pathologic result as squamous cell carcinoma.
* Neurological or mental abnormalities which affect cognitive ability.
* Severe cardiovascular and cerebrovascular diseases, such as heart failure (NYHA III-IV class), uncontrolled coronary heart disease, cardiomyopathy, uncontrolled arrhythmias, uncontrolled hypertension, myocardial infarction or cerebral infarction within past six months.
* Active serious clinical infections :> Class 2 NCI-Common Toxicity Criteria for Adverse Effects (CTCAE) Version 4.0 within 14 days before randomization, including active tuberculosis.
* HIV infection or active hepatitis B or hepatitis C.
* Uncontrolled systemic diseases, such as poorly controlled diabetes mellitus.
* Medical history of interstitial lung disease, such as interstitial pneumonia, pulmonary fibrosis, or baseline chest X-ray / CT showed evidence of interstitial lung disease;
* Pregnancy (via urine β-human chorionic gonadotropin test to determine) or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
local control rate | 1 year
  According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 standard, tumor progressing during the treatment and follow up period means local control failure, which include the sum of diameters of local and region target focus increases ≥20% or ≥5mm; new focus emerges at local or region area; metastases or secondary primary tumor would not be concluded.

SECONDARY OUTCOMES:
progression-free survival | 2 years
  progression-free survival is definite as the time of death of tumor progression event emerges from the patient was randomize. According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 standard, tumor progressing during the treatment and follow up period means local control failure, which include the sum of diameters of local and region target focus increases ≥20% or ≥5mm; new focus emerges at local or region area; metastases or secondary primary tumor would not be concluded. No respondent means the tumor advances at the first day.
overall survival | From date of randomization until the date of death from any cause, assessed up to 2 years
  Refers to the result from a random start time to death of any cause. Records from the beginning of the random time to time of any cause of death. Shedding of subjects censored cases recorded censored time.

OTHER OUTCOMES:
quality of life | 2 year
  Measured using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Scale Quality of life Questionnaire (QLQ)-C30 (V3.0) and the QLQ-H & N35 (V1.0) of quality of life questionnaire.
The incidence of radiation-related adverse reactions | 2 years
  according to NCI-Common Toxicity Criteria Adverse Event （CTCAE）4.0 standard

CONTACTS AND LOCATIONS:
Overall Officials: Jianguo Zhang, Doctor, Study Director — Peking University, School of Stomatolgy; Yan Sun, Doctor, Principal Investigator — Peking Univesity, Beijing Cancer Hospital
Locations (1):
- Peking University, School and Hospital of Stomatology, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu SM, Wang HB, Sun Y, Shi Y, Zhang J, Huang MW, Zheng L, Lv XM, Zheng BM, Reilly KH, Yan XY, Ji P, Wu YF, Zhang JG. The efficacy of iodine-125 permanent brachytherapy versus intensity-modulated radiation for inoperable salivary gland malignancies: study protocol of a randomised controlled trial. BMC Cancer. 2016 Mar 7;16:193. doi: 10.1186/s12885-016-2248-7. PMID 26951097